CLINICAL TRIAL: NCT01760213
Title: Internet Based Treatment Using Virtual Reality in the Prevention of PTSD
Brief Title: Brief Internet Based Treatment for PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: VRInternet
Record Dates: First submitted 2012-12-12; First posted 2013-01-04 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2012-12

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): intervention delivered via internet
  Interventions: Other: CBT delivered via Internet
- Control (No Intervention)

INTERVENTIONS:
Other: CBT delivered via Internet
  Arms: Treatment

SUMMARY:
The goal of the project is to overcome some of the common barriers to treatment amongst recent survivors of traumatic events, by combining the world of evidence-based intervention with that of modern Internet technology. Specifically, it aims to test the feasibility and effectiveness of an Internet delivery of early-intervention trauma-focused cognitive behavioral therapy (CBT) for preventing post-traumatic stress disorder (PTSD). Over the course of the study the following objectives will be achieved:

1. The development of an Internet-based Virtual Reality intervention for preventing PTSD among patients who have recently experienced a traumatic event.
2. The evaluation of the feasibility of administering this intervention, and
3. The evaluation of the efficacy of this Internet based intervention in the prevention of PTSD in recent trauma survivors.

ELIGIBILITY:
Inclusion Criteria:

* Exposed to a traumatic event that meets DSM Criteria (objectively could cause physical injury;
* Subjectively involves helplessness or fear);
* Aged over 18; Aged under 65;
* Hebrew speaking; Suffering from PTSD (without the time criteria i.e. less than one month of symptoms);
* Able to give informed consent.

Exclusion Criteria:

* Suffering from, or have suffered from in the past, bipolar disorder;
* Suffering from, or have suffered from in the past, psychotic disorder;
* Suffering from, or have suffered from in the past, substance abuse;
* Suffering from PTSD;
* Suffering from another Axis I anxiety disorder that requires immediate treatment;
* Currently presents as a suicide risk, requiring hospitalization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Levels of PTSD symptoms | 12 months after end of treatment
  the main outcome measure will be PTSD symptoms as measured by the CAPS.

CONTACTS AND LOCATIONS:
Overall Officials: Rena Cooper, MD, Principal Investigator — HMO; Sara Freedman, PhD, Study Director — Bar Ilan University
Locations (1):
- Hadassah medical organization, Jerusalem, Israel, Israel